CLINICAL TRIAL: NCT03089671
Title: Optimal Ureteric Visualization At the Time of Pelvic Reconstructive Surgery: Vitamin B Versus 5% Dextrose in Water
Brief Title: Ureteric Visualization: Vitamin B Vs 5% Dextrose in Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FPMRS McD 001
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Pelvic Floor Disorders; Ureter; Kink
Keywords: Vitamin B; 5% Dextrose in Water; Cystoscopy; Ureter
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Folic Acid; Riboflavin; Glucose; Water

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Patient packages will be created and assigned a kit number. For those randomized to the vitamin B2 group, the package will consist of a pill of vitamin B2 (100mg riboflavin) inside an opaque gelatin capsule that is matched to a litre bag of normal saline wrapped in an opaque covering. For those randomized to the D5W group, the package will consist of a pill that is a placebo pill (opaque gelatin capsule of microcrystalline cellulose powder) matched to a litre bag of D5W wrapped in an opaque covering. These packages will be coupled with the patient according to her randomization group in the preoperative area.
  In the preoperative area, all patients will be given the pill in their package by mouth 60 to 120 minutes before the start of surgery. The covered bag will then accompany the patient to the operating room and will be set up as the instillation fluid for cystoscopy. This way, the patient and operating team will be blinded to the agent used for ureteric visualization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B (Experimental): Vitamin B: Patients in this arm will receive 100mg of riboflavin (vitamin B2) 60 to 120 minutes prior to surgery for the purpose of turning the urine bright yellow to see if this helps with detection of ureteric jets during cystoscopy which will be done using normal saline.
  Interventions: Other: Vitamin B (riboflavin, vitamin B2)
- D5W (5% dextrose in water) (Active Comparator): 5% Dextrose in Water: Patients in this arm will receive a placebo in the pre-operative area (for the purpose of blinding the surgical team) 60 to 120 minutes prior to surgery. Intraoperative cystoscopy will then be performed using D5W to see if this helps with detection of ureteric jets.
  Interventions: Other: 5% Dextrose in Water (D5W)

INTERVENTIONS:
Other: Vitamin B (riboflavin, vitamin B2) — Vitamin B is a natural health product approved as a colouring agent.
  Arms: Vitamin B
Other: 5% Dextrose in Water (D5W) — 5% Dextrose in Water is an irrigation/instillation fluid, commonly used in intravenous lines.
  Arms: D5W (5% dextrose in water)

SUMMARY:
Background: The risk of ureteric injury at the time of pelvic reconstructive surgery can be as high as 3% and the American College of Obstetricians and Gynecologists has stated that intraoperative cystoscopy should be done after all such procedures. Intravenous indigo carmine was routinely given during surgery to colour the urine bright blue and allow for assessment of ureteric integrity. In 2014, indigo carmine was no longer available worldwide and since then, surgeons have been searching for suitable alternatives. Vitamin B is a water soluble vitamin that colours the urine bright yellow and can be given immediately before surgery to help with ureteric visualization. Alternatively, 5% dextrose in water (D5W) can be used as the instillation fluid during cystoscopy to allow for urine jet visualization due to the difference in fluid viscosity. Both agents have been shown to be better than instillation with normal saline and are affordable and accessible in Canada.

Objective: To identify which agent is superior for intraoperative ureteric visualization at the time of cystoscopy by determining the difference in detection rate of both ureteric jets using either preoperative oral vitamin B or intraoperative cystoscopic distension with D5W.

Methods: This study will be a three-site (Mount Sinai Hospital, Sunnybrook Health Sciences Centre, Women's College Hospital), double-blinded, randomized control trial whereby female patients undergoing pelvic reconstructive surgery will be randomized to receive either preoperative vitamin B or intraoperative D5W cystoscopic instillation fluid. Parameters measured during surgery will include whether both ureteric jets were seen, time to visualization of both ureters, colour of jets, and surgeon satisfaction. Patients will also be seen at one week after surgery to assess for urinary tract infection. Sample size calculation based on previous studies demonstrated a need for 119 patients per study arm.

Anticipated Clinical Significance: The findings of this study will be relevant to all surgeons performing intraoperative cystoscopy where ureteric visualization is required. The investigators believe the outcome of this study will help make cystoscopy shorter and more efficient for surgeons who often feel the pressure of time constraints within the operating room setting. In turn, decreasing the time of cystoscopy may reduce operating times which will benefit both the patient and hospital.

DETAILED DESCRIPTION:
Study Design: This study will be a double blinded, randomized control trial (RCT) to compare detection rates of one and both ureteric jets at the time of intraoperative cystoscopy using either vitamin B or D5W. This will be a multicentre study with patients being recruited from Mount Sinai Hospital, Sunnybrook Health Sciences Centre, and Women's College Hospital.

Recruitment and Consent: Female patients undergoing pelvic reconstructive surgery where cystoscopic ureteric visualization is required will be recruited from Mount Sinai Hospital/Sunnybrook Health Sciences Centre/Women's College Hospital at their surgical consult in the clinic/ambulatory setting. At that time, one of the study investigators (not the operating physician for that particular patient) will describe the study to the patient and give her the study consent form if she is interested in participating. For any patients recruited or considering the study, they will be asked to stop all vitamin supplements one week before surgery. If the patient cannot decide on the day of the surgical consult, they can go home with an unsigned consent form to review the study and on the day of surgery they will once again be asked if they would like to participate in the study by a study investigator (not involved with the patient's surgery). Once the patient has read and voluntarily signed the consent form, the same study investigator will open a sequentially numbered opaque sealed envelope that will provide a study identification number for the patient and randomize the patient to either receiving a preoperative dose of vitamin B or intraoperative cystoscopic distension with D5W. The patient and operating surgeons will not be made aware of the group the patient was allocated to.

Sample Size Calculation: There is only one study in the literature that has commented on ureteric visualization after vitamin B2 ingestion. In this study, they report a 72% detection rate. If we consider a 15% difference in detection rate to be clinically significant, then with a power of 0.8 and an alpha of 0.05, the minimum number of patients required per group would be 113. We anticipate a 5% drop out rate after consent due to intraoperative issues. Therefore, we will recruit 119 patients per study arm to be included in the final analyses (n=238).

Method: Upon recruitment to the study, the study investigator that did the consent will then complete the Initial Information Form where the following information will be collected from the patient (this information is also already available in the clinical record):

* Age
* Parity
* BMI
* Smoking status
* Diabetic status
* Menopausal status
* Immunocompromised status
* Pelvic Organ Prolapse-Quantification (POP-Q) stage
* Preoperative use of vaginal estrogen
* History of recurrent UTI

Patient packages will be created and assigned a patient number. For those randomized to the vitamin B group, the package will consist of a pill of vitamin B2 (containing 100mg of riboflavin) that is inside an opaque gelatin capsule that is matched to a litre bag of normal saline that is wrapped in an opaque covering. For those randomized to the D5W group, the package will consist of a pill of cellulose that is inside an opaque gelatin capsule that is matched to a litre bag of D5W that is wrapped in an opaque covering. These packages will be couple with the patient according to her randomization group in the preoperative area.

In the preoperative area, all patients will be given the pill in their package by mouth 60 to 120 minutes before the start of surgery. The covered bag will then accompany the patient to the operating room and will be set up as the instillation fluid for cystoscopy. This way, the patient and operating team will be blinded to what agent was used for ureteric visualization. Cystoscopy will be done using a standard diagnostic 70 degree cystoscope.

In the preoperative area and in the operating room, the following data will be collected by a study investigator that is not part of the operating team:

* Time pill was given
* Time cystoscopy was started
* Time surgeon started to look for ureteric jets
* Time first ureter was visualized
* Time second ureter was visualized
* Colour of jet (clear, pale yellow, or bright yellow)
* If cystoscopy is repeated to look at ureters, above measures are captured again
* If fluorescein (0.25mL by iv injection) is used as a rescue agent, reason why, time it was given, and time jets were seen are recorded (in order to allow for an adequate time to determine whether the study agent has worked, fluorescein cannot be used any earlier than 10 minutes from the start of cystoscopy)
* Surgeon satisfaction of ureteric visualization during that specific case is rated on a Likert scale from 1 to 5
* Primary surgeon's guess at the agent that was used to visualize ureters

Between post-operative days 3 and 10, the patient will present to clinic and information on length and type of catheter use, as well as antibiotic use after surgery will be recorded. Patients will also give a catheter urine specimen to be sent for culture and sensitivity.

DATA ANALYSIS Baseline characteristics and follow-up measures will be summarized using descriptive statistics (mean, SD, median, and range for continuous variables, count and percent for categorical variables). Continuous variables will be summarized using means and standard deviations, and will be compared between groups using Student's t-tests. Categorical variables will be summarized using counts and percents, and compared between groups using Chi-squared tests. A P-value ≤0.05 will be considered significant for all statistical analyses performed.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing pelvic reconstructive surgery for pelvic organ prolapse where cystoscopy is necessary to assess ureteric integrity

Exclusion Criteria:

* Known kidney disease
* Known ureteral disease or previous ureteric compromise
* Patients with known hypersensitivity to cyanocobalamin or cobalt
* Known malabsorption disorder
* Known allergy to fluorescein dye
* Unable to present for one week post-operative assessment due to geographic or transportation issues
* Unable to provide written consent to the study as a result of language barriers or cognitive disabilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients recruited for the study will be undergoing female pelvic floor surgery.
Enrollment: 238 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Detection rates of both ureteric jets at the time of intraoperative cystoscopy using either preoperative oral vitamin B or intraoperative distension with D5W. | If ten minutes has passed and no jets are seen the surgeon is allowed to ask for iv fluorescein for visualization and this would be considered a failed detection.
  Visual queue: detection will be counted as occurring when both ureteric jets are seen

SECONDARY OUTCOMES:
Difference in time to visualization of one and both ureters using either preoperative oral vitamin B or intraoperative cystoscopic distension with D5W. | Time will be measured from the time the surgeon states they have started looking for ureteric jets to the time that one and both ureteric jets are seen. This time period will be up to ten minutes.
  Time assessment
Difference in the number of times intravenous fluorescein is used as a rescue agent to visualize ureters when vitamin B or D5W has failed. | Number of times fluorescein is used during intraoperative cystoscopy to visualize ureters when experimental agents have failed.
  Count
Difference in surgeon satisfaction when using vitamin B or D5W. | Done after surgery is complete in the operating room
  Visual analog satisfaction scale
Difference in urinary tract infection rates after surgery after using vitamin B or D5W. | Urine will be collected 3 to 10 days after surgery.
  Infection rates

CONTACTS AND LOCATIONS:
Overall Officials: Colleen D McDermott, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers